CLINICAL TRIAL: NCT04781075
Title: TAP (Transverse Abdominis Plane) Block With Exparel (Liposomal Bupivicaine) vs. Bupivicaine Post-op Pain Management
Brief Title: Modified TAP (Transverse Abdominis Plane) Block in Colorectal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ochsner Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017.044 -TAP Block
Record Dates: First submitted 2019-04-11; First posted 2021-03-04 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- TAP Block with Exparel (Experimental): TAP Block with 20 mL (266mg) of liposomal bupivacaine with 25 mL (5 mg/mL) of bupivacaine diluted in 55 mL of normal saline
  Interventions: Other: Pain Scale; Drug: Exparel Injectable Product
- TAP Block with bupivicaine (Active Comparator): TAP Block with 30 mL (5mg/mL) of bupivacaine diluted in 70 mL of normal saline
  Interventions: Other: Pain Scale; Drug: Bupivacaine Injection

INTERVENTIONS:
Other: Pain Scale — Maximum Daily Pain Scale will be recorded daily until discharge (typically under 7 days)
Drug: Exparel Injectable Product — Given at the beginning of the surgery for post-operative pain management
  Arms: TAP Block with Exparel
Drug: Bupivacaine Injection — Given at the beginning of the surgery for post-operative pain management
  Arms: TAP Block with bupivicaine

SUMMARY:
Single Blind, Randomized Controlled study to see if TAP Block with Exparel provides better pain relief than TAP Block with bupivicaine. Differences in Pain Scale, Length of Stay, and Total Narcotic use in the hospital will be evaluated.

DETAILED DESCRIPTION:
Subjects recruited into the study will undergo surgery as scheduled. During the procedure they will receive a TAP Block with one of the pain medications. TAP Block in the experimental arm will be performed with 20 mL (266mg) of liposomal bupivacaine with 25 mL (5 mg/mL) of bupivacaine diluted in 55 mL of normal saline. The control arm will have a TAP Block performed with 30 mL (5mg/mL) of bupivacaine diluted in 70 mL of normal saline. These doses are consistent with prior studies of TAP Block with liposomal bupivacaine. Subjects will be monitored for pain as per standard of care and will be given pain medication as needed.

Subject Recruitment and Screening Patients will be recruited from the Ochsner Colorectal Surgery Clinic at the time of a preoperative visit.

Study Procedures

Screening & Baseline Visit After obtaining informed consent the subjects relevant medical and surgical history will be documented. Demographics and vitals will be documented. Current use of pain medication will be recorded. A physical exam will be performed.

Day of Surgery Routine vital signs will be obtained preoperatively. During the operation subject will receive a TAP Block containing their randomized local injection mixture as described above. Following surgery the subject will recover the PACU and pain medication will be provided on demand. Initial postoperative vital signs and pain scores will be obtained at this time.

Post-Operative Course Postoperatively subject will have regularly scheduled vital signs and pain scores obtained, and recorded for study use. Narcotic and non-narcotic pain medication will be provided on demand; dosages will be recorded for study use. Subjects will be followed until they are discharged at which time study participation will be complete.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18-75 years undergoing planned laparoscopic colon or rectal resection

Exclusion Criteria:

1. Patients younger than 18 or older than 75 years old
2. Pregnant women
3. Patients who have taken steroids or other immunomodulators within the last 6 months
4. Patients on home narcotics
5. Patients allergic to Exparel or bupivacaine

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Pain Scale | daily through study completion (up to 30 days)
  Daily Pain Scale using Wong-baker FACES Pain Rating Scale 0 (no pain) - 10 (worst pain imaginable)

SECONDARY OUTCOMES:
Length of stay | daily through study completion (up to 30 days)
  Duration of hospitalization post-operatively
Narcotic use | daily through study completion (up to 30 days)
  Total amount of narcotic used for pain control postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Charles Whitlow, MD, Principal Investigator — Ochsner
Locations (1):
- Ochsner Medical Center, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chevrollier GS, Klinger AL, Green HJ, Gastanaduy MM, Johnston WF, Vargas HD, Kann BR, Whitlow CB, Paruch JL. Liposomal Bupivacaine Transversus Abdominis Plane Blocks in Laparoscopic Colorectal Resections: A Single-Institution Randomized Controlled Trial. Dis Colon Rectum. 2023 Feb 1;66(2):322-330. doi: 10.1097/DCR.0000000000002346. Epub 2022 May 24. PMID 35849756